CLINICAL TRIAL: NCT00721864
Title: The Molecular Biology of Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Josef T. Prchal, MD, University of Utah
Other Study IDs: 17790; R01HL5077-12
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Hemoglobinuria, Paroxysmal
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PIG-A Mutation; Prion Protein; Hematopoietic stem cells; Clonal disorder
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Insomnia, Fatal Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Affected Population: Subjects suspected of having Paroxysmal Nocturnal Hemoglobinuria (PNH)

SUMMARY:
This study is designed to better understand the molecular biology of paroxysmal nocturnal hemoglobinuria (PNH) and to determine if prion protein (PrP) functions in long term hematopoietic stem cell renewal.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is characterized by hemolytic anemia, thrombosis, and variable cytopenia. It can be associated with significant morbidity including acute kidney failure, cerebral infarction, mesenteric infarction, Budd-Chiari syndrome, aplastic anemia, and leukemic transformation. The average survival time from diagnosis is 15 years.

PNH is an acquired clonal disorder of the hematopoietic stem cell. Two distinct populations of hematopoietic cells exist in each PNH patient: one non-clonal population of normal cells, and one clonal population of PNH cells. The clonal population of PNH cells is identified by a mutation in the PIG-A gene that results in absence of the glycophosphatidylinositol (GPI) anchor of several surface proteins. Consequently, these surface proteins are unable to perform their functions on the cell surface. Deficiency of two of these surface proteins, CD55 (decay accelerating factor) and CD59 (membrane inhibitor of reactive lysis) that prevent complement mediated destruction, have been shown to underlie the clinical presentation of PNH. Identifying the mutation causing the predominant clones may help us better understand the molecular biology of PNH. When this is accomplished, new therapies to control and eventually cure the disease can be designed.

In addition, we propose to determine the function of PrP in human hematopoietic stem cells. PrP is a glycoprotein attached to the cell membrane by a glycosylphosphatidylinositol (GPI) anchor. In PNH, a disorder whose pathogenesis lies in the absence of GPI anchors, PrP expression is reduced in monocytes and granulocytes from the PNH clone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects suspected of or diagnosed with Paroxysmal Nocturnal Hemoglobinuria (PNH)
2. Age > 7

Exclusion Criteria:

1. Those not meeting the inclusion criteria

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with paroxysmal nocturnal hemoglobinuria (PNH)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Identify the mutation causing the predominant clones through analysis of extracted DNA/RNA from erythroid colonies | After sample is obtained

SECONDARY OUTCOMES:
Reconfirmation of PrP expression in human granulocytes, hematopoietic progenitors and stem cells | After sample is obtained
Analysis of PrP function in human long term hematopoietic stem cells | After sample is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Durig J, Giese A, Schmucker U, Kretzschmar HA, Duhrsen U. Decreased prion protein expression in human peripheral blood leucocytes from patients with paroxysmal nocturnal haemoglobinuria. Br J Haematol. 2001 Mar;112(3):658-62. doi: 10.1046/j.1365-2141.2001.02602.x. PMID 11260069
- [Background] Risitano AM, Holada K, Chen G, Simak J, Vostal JG, Young NS, Maciejewski JP. CD34+ cells from paroxysmal nocturnal hemoglobinuria (PNH) patients are deficient in surface expression of cellular prion protein (PrPc). Exp Hematol. 2003 Jan;31(1):65-72. doi: 10.1016/s0301-472x(02)01011-1. PMID 12543108
- [Background] Zhang CC, Steele AD, Lindquist S, Lodish HF. Prion protein is expressed on long-term repopulating hematopoietic stem cells and is important for their self-renewal. Proc Natl Acad Sci U S A. 2006 Feb 14;103(7):2184-9. doi: 10.1073/pnas.0510577103. Epub 2006 Feb 7. PMID 16467153